CLINICAL TRIAL: NCT05923736
Title: Assessment of Cardiovascular Risk in Digital Osteoarthritis: A Case-control Study.
Brief Title: Cardiovascular Risk in Digital Osteoarthritis
Acronym: RICARDI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AOI 2022 MATHIEU
Record Dates: First submitted 2023-06-15; First posted 2023-06-28 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2023-04

CONDITIONS: Osteoarthritis Hand; Lumbago; Osteoporosis; Radiculopathy Lumbar
MeSH Terms: conditions — Low Back Pain; Osteoporosis | interventions — Absorptiometry, Photon

STUDY DESIGN:
Intervention Model Description: It's a cross-sectional case-control study. The study will include patients with digital osteoarthritis as case group and patients with lumbago and osteoporosis without a inflammatory arthritis as control group.Imaging exams will be added for research purposes, and are not part of routine care or diagnosis of these conditions: intima-media thickness, arterial compliance and arterial composition; these tests involve minimal risk.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Case group : digital osteoarthritis (Other)
  Interventions: Other: Intima media thickness ultrasound; Other: hand ultrasound; Other: EndoPAT™ 2000 system; Other: X-ray absorptiometry (DXA)
- Control group : lumbago, osteoporosis (Other)
  Interventions: Other: Intima media thickness ultrasound; Other: hand ultrasound; Other: EndoPAT™ 2000 system; Other: X-ray absorptiometry (DXA)

INTERVENTIONS:
Other: Intima media thickness ultrasound — EIM is a non-invasive ultrasound technique in which an ultrasound-generating probe is conventionally placed opposite the right primary carotid artery. By distinguishing between an inner layer, consisting of the intima and media, and the outer layer, the adventitia, the intima-media thickness can be assessed.
Other: hand ultrasound — Performed by the rheumatologist, to quantify the number of synovial thickenings in B mode and the number of synovitis in Doppler mode. The presence or absence of joint erosions on the metacarpophalangeal (MCP), proximal interphalangeal (PPI) or distal interphalangeal (DIP) joints.
Other: EndoPAT™ 2000 system — It's a measurement that detects endothelial dysfunction in coronary arteries using reactive hyperemia.This examination will be carried out in accordance with the manufacturer's instructions by the Rheumatology Department nurse. The patient lies down for the duration of the examination (20 minutes). A probe is placed on the index finger of each hand and a cuff on the left arm. Recording begins with a 5-minute baseline period (at rest), followed by a 5-minute period of arm occlusion, and ends with a 5-minute period of return to normal.
Other: X-ray absorptiometry (DXA) — This X-ray examination will be carried out on the Hologic device and the analyses by APEX 4.0 software. Two-photon X-ray absorptiometry (DXA) is a method commonly used to measure bone mineral density. It is based on a scan of the body by an X-ray beam at 2 different energy levels, which enables 3 compartments to be individualized: mineral mass, lean mass and fat mass. This low-radiation method (less than a conventional chest X-ray) is regarded as a benchmark for accurate measurement of both bone mineral density and the various body compartments. The examination lasts 10 minutes and is carried out by the department's electroradiology manipulators

SUMMARY:
The goal of this cross-sectional case control study is to investigate the cardiovascular risk in digital osteoarthritis. This study aims to compare the cardiovascular risk between group of patients with digital osteoarthritis and control group of patients with non-osteoarthritis disease paired by measurement of carotid intima-media thickness. All participants will undergo an ultrasound scan to measure carotid intima media thickness, a clinical assessment with the rheumatologist and a cardiovascular risk assessment.

ELIGIBILITY:
Inclusion Criteria:

For all subjects:

* Adult male or female subject
* Able to give informed consent to participate in research
* Affiliated with a Social Security plan

For the digital osteoarthritis group:

* Consultant in Rheumatology at Clermont-Ferrand University Hospital
* Affected by digital osteoarthritis meeting ACR diagnostic criteria with radiographic signs of osteoarthritis validated by a radiologist.

For the control group :

* Rheumatology consultant at the Clermont-Ferrand University Hospital or hospitalized in this department for a non-arthritic, non-rheumatic pathology.
* Patients with spinal disc pathology (lumbago, radiculalgia due to disco-radicular conflict) or non-severe osteoporosis, i.e. with a densitometric T score between -2.5 and -3 DS.

Exclusion Criteria:

For all topics :

* Refusal to participate
* Pregnant women, nursing mothers
* Subjects under guardianship or curatorship, deprived of liberty, or under court protection

For the digital osteoarthritis group:

- Existence of diagnostic arguments for another inflammatory rheumatism (rheumatoid arthritis, spondylarthritis, psoriatic arthritis, lupus, gout, chondrocalcinosis...) or another arthrosic localization (gonarthrosis, coxarthrosis, discarthrosis) symptomatic at the time of inclusion or affecting daily activities.

For the control group :

* Existence of chronic inflammatory rheumatism (rheumatoid arthritis, spondylitis, psoriatic arthritis, lupus, gout, chondrocalcinosis...)
* Existence of digital osteoarthritis
* Existence of another painful arthritic site (knee, hip, rachi) Existence of finger pain, whatever the etiology.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-10-04 (Actual); Primary Completion 2025-10-04 (Estimated); Study Completion 2026-10-04 (Estimated)

PRIMARY OUTCOMES:
Measurement of carotid intima-media thickness | 20 minutes
  EIM is a non-invasive ultrasound technique in which an ultrasound-generating probe is conventionally placed opposite the right primitive carotid artery. By distinguishing between an inner layer, consisting of the intima and media, and the outer layer, the adventitia, the intima-media thickness can be assessed.

SECONDARY OUTCOMES:
Cardiovascular risk assessment by SCORE scale | 10 minutes
  The SCORE scale measures the percent risk of a fatal cardiovascular event at 10 years due to arteriosclerosis.
Identify endothelial dysfunction in coronary arteries by reactive hyperemia index score | 15 minutes
  The EndoPAT™ 2000 device (Itamar medical) is an examination to detect endothelial dysfunction in coronary arteries using reactive hyperemia: Normal EndoScore™: RHI > 1.67; Abnormal EndoScore™: RHI ≤ 1.67 .
Measurement of bone mineral density and body mass composition by DXA | 15 minutes
  Two-photon X-ray absorptiometry (DXA) is a method commonly used to measure bone density. The examination distinguishes between 3 measurements: mineral mass, lean mass and fat mass.
Physical performance assessment by measuring the distance covered in metres in 6 minutes over a 30-metre course | 6 minutes
  Patients walk in a rhythmic sequence for 6 minutes on a 30-metre distance,this assesses the muscular strength of the lower limbs and enables you to judge your physical level

CONTACTS AND LOCATIONS:
Overall Officials: Sylvain Mathieu, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Chu Clermont Ferrand, Clermont-Ferrand, France